CLINICAL TRIAL: NCT00379093
Title: Preventing Harm From Alcohol Use in Older Adults
Brief Title: Healthy Living as You Age
Acronym: HLAYA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Alison A. Moore, MD, MPH - Principal Investigator, University of California, Los Angeles, David Geffen School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIAAA-MOO-013937; NIH Grant 5 RO1 AA 013937
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Alcohol Related Disorders; Alcohol Drug Interactions
Keywords: Alcohol; Comorbidity; Aging; Brief Advice; Randomized Trial
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Brief advice — The intervention will have the following components:
  A) At the time of the recruitment visit, all intervention group patients will receive:
  * A personalized risk report;
  * An educational booklet titled "Healthy Drinking as You Age";
  * A drinking diary;
  * Brief advice to reduce their drinking by their physicians;
  B) After the recruitment visit, all intervention group patients will receive up to 3 telephone calls from a health educator. After each call, intervention group patients may choose to receive a letter updating their health risks.
  Also, at the conclusion of their interaction with the health educator, they may choose to have a letter summarizing the calls sent to their physician.

SUMMARY:
Older persons who drink can be vulnerable to negative consequences of drinking. This trial aims to prevent harm from alcohol use in older adults through a program of screening and brief advice followed up with several health education phone calls.

DETAILED DESCRIPTION:
Approximately 50% of persons aged 65 years and older drink alcohol. Older persons are particularly susceptible to adverse consequences of drinking such as falls, depression, sleep disorders, stomach upset, hypertension, and alcohol/drug interactions. This is because of age-related changes in the body that affect how older persons react to alcohol and also because of the age-associated increases in illness and medication use.

In the current project we aim to see if screening and brief advice given to older risky drinkers in a physician's office followed by up to 3 health education phone calls may reduce their risks associated with alcohol use. We plan to use a newly developed and tested measure, the Comorbidity Alcohol Risk Evaluation Tool (CARET), to screen for older persons (aged 55 and older) whose use of alcohol alone or in combination with their illnesses, symptoms, and medication use may be causing them harm, or increasing their risk for harm. Persons whose responses on the CARET indicate they might be risky drinkers will be randomized to receive either a brief intervention to reduce their risks or usual care.

The intervention will have the following components:

A) At the time of the recruitment visit, all intervention group patients will receive:

1. A personalized risk report;
2. An educational booklet titled "Healthy Drinking as You Age";
3. A drinking diary;
4. Brief advice to reduce their drinking by their physicians;

B) After the recruitment visit, all intervention group patients will receive up to 3 telephone calls from a health educator. After each call, intervention group patients may choose to receive a letter updating their health risks. Also, at the conclusion of their interaction with the health educator, they may choose to have a letter summarizing the calls sent to their physician.

At the time of the recruitment visit, control group patients will receive a booklet on a variety of healthy behaviors titled "Healthy Living as You Age." Both control and intervention group patients will receive a telephone call from a research associate 3 months and 12 months after initial enrollment in the study to administer the CARET again.

We will analyze our results to look for differences between the intervention and control groups at 12 months in the a) proportions of them identified as risky drinkers by the CARET; b) the amount they drink; c) the numbers of risks identifying those persons who are still risky drinkers and d) the difference in their expectations regarding aging.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years of age
* Seeing a participating physician (internists or family physicians employed at any of the participating sites)
* Have had at least one alcoholic drink in the last week

Exclusion Criteria:

* Too ill to participate
* Have received substance abuse services in past 3 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2003-08; Primary Completion 2007-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Reducing at-risk drinking | 12 month

SECONDARY OUTCOMES:
Reducing alcohol use | 12 month
Reducing the number of risks among those still considered at-risk drinkers. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Alison A. Moore, MD, MPH, Principal Investigator — UCLA DOM-Geriatrics
Locations (1):
- UCLA Department of Medicine, Geriatrics Research Center, Los Angeles, California, United States